CLINICAL TRIAL: NCT02767297
Title: A Three-Part Phase 1b Bioavailability and Pharmacokinetics Study of Two Formulations of FDL169 in Healthy Subjects and Subjects With Cystic Fibrosis
Brief Title: Bioavailability and Pharmacokinetics Study of FDL169 in Healthy Subjects and Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Flatley Discovery Lab LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: FDL169-2015-03
Record Dates: First submitted 2016-05-05; First posted 2016-05-10 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1: Single dose (cross over) (Experimental): FDL169 reference formulation and test formulation administered as a single dose in healthy subjects
  Interventions: Drug: FDL169
- Part 2: Multiple dose (dose level 1) (Experimental): FDL169 test formulation (Dose level 1) administered as repeat doses in healthy subjects
  Interventions: Drug: FDL169
- Part 2: Multiple dose (dose level 2) (Experimental): FDL169 test formulation (Dose level 2) administered as repeat doses in healthy subjects
  Interventions: Drug: FDL169
- Part 2: Multiple dose (dose level 3) (Experimental): FDL169 test formulation (Dose level 3) administered as repeat doses in healthy subjects
  Interventions: Drug: FDL169
- Part 3: Single dose (Experimental): FDL169 test formulation administered as a single dose in CF subjects
  Interventions: Drug: FDL169

INTERVENTIONS:
Drug: FDL169

SUMMARY:
To determine the relative bioavailability of the capsule (reference) and tablet (test) formulations of FDL169 in healthy adult males and females, and to evaluate the pharmacokinetic (PK) profile FDL169 tablets (test formulation) in both healthy adult males and females, and subjects with cystic fibrosis (CF).

DETAILED DESCRIPTION:
This is a three-part study.

Part 1:

Part 1 of the study is a single dose, open-label, randomized crossover study in healthy male and female subjects to compare the relative bioavailability of two formulations of FDL169.

Part 2:

Part 2 of the study is a multiple, escalating dose study of three different doses of the test formulation of FDL169 in healthy male and female subjects to evaluate the PK profile of the test formulation of FDL169.

Part 3:

Part 3 of the study is a single dose, open-label study in male and female subjects with CF to determine the PK profile of the test formulation of FDL169.

ELIGIBILITY:
Inclusion Criteria:

Parts 1 and 2:

1. Healthy, males and females between 18 and 55 years of age, inclusive, with a BMI of >19 and <30 kg/m2.
2. If sexually active, must meet the contraception requirements.

Part 3:

1. Male and female subjects aged 18 years and older.
2. If sexually active, must meet the contraception requirements.
3. Diagnosis of CF.
4. History of pancreatic insufficiency.
5. Forced expiratory volume in 1 second (FEV1) ≥40% of predicted normal for age, sex and height at screening.

Exclusion Criteria:

Parts 1 and 2:

1. Prior or ongoing medical condition, medical history, physical findings, ECG findings or laboratory abnormality that could adversely affect the safety of the subject.
2. Alkaline phosphatase, aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) level >1.5 x upper limit of normal (ULN) at screening.
3. Use of prescription or non-prescription drugs within 21 days or five half-lives (whichever is longer) before the first dose of study medication, unless the medication will not interfere with the study procedures or compromise subject safety.
4. Pregnant or nursing females.
5. Serum creatinine or total bilirubin >1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).
6. History of prolonged QT and/or QTcF interval.
7. ECG with a single QTcF >450 msec in males, >460 msec in females, at Screening.
8. Positive urinary drugs of abuse screen at Screening or Day -1, or positive alcohol screen at Day -1.
9. History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units.
10. History of human immunodeficiency virus (HIV) or positive HIV, hepatitis B or hepatitis C results at screening.
11. Donation of 500 mL or more blood within 3 months before Day -1.
12. Participation in a clinical trial involving receipt of an investigational product within the past 90 days or exposure to more than four new chemical entities with 12 months of the first dosing day.
13. Current smoking or use of tobacco products or substitutes. Former smokers will be eligible, provided they have not smoked for at least 6 months before Day -1.
14. Use of any prescription and non-prescription medications that are inhibitors or inducers of cytochrome P450 (CYP) 3A4 within 7 days before Day -1.

Part 3:

1. History of any illness, or ongoing acute illness that could impact the safety of the subject or confound study results.
2. Abnormal liver function ≥3 x ULN: AST, ALT, total bilirubin.
3. A pulmonary exacerbation, or changes in therapy for pulmonary disease within 4 weeks prior to the Baseline (Day 1) Visit
4. Use of herbal and dietary supplements within 21 days or five half-lives (whichever is longer) before the first dose of study medication, unless the medication will not interfere with the study procedures or compromise subject safety.
5. Pregnant or nursing females.
6. Serum creatinine or total bilirubin >1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).
7. History of prolonged QT and/or QTcF interval.
8. ECG with a single QTcF >450 msec in males, >460 msec in females, at Screening.
9. Positive urinary drugs of abuse screen at Screening or Day -1, or positive alcohol screen at Day -1.
10. History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units.
11. History of HIV, or positive HIV, hepatitis B or hepatitis C results at screening.
12. Donation of 500 mL or more blood within 3 months before Day -1.
13. Participation in a clinical trial involving receipt of an investigational product within the past 90 days or exposure to more than four new chemical entities with 12 months of the first dosing day.
14. Current smoking or use of tobacco products or substitutes. Former smokers will be eligible, provided they have not smoked for at least 6 months before Day -1.
15. Use of any prescription and non-prescription medications that are inhibitors or inducers of CYP3A4, within 7 days before Day -1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum plasma concentration of FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 72 h post-dose
Part 1: Time to maximum plasma concentration of FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 72 h post-dose
Part 1: Individual estimate of the terminal elimination rate constant of FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 72 h post-dose
Part 1: Terminal half-life of FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 72 h post-dose
Part 1: AUC from the time of dosing to the time of the last observed concentration for FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 72 h post-dose
Part 1: AUC extrapolated to infinity from dosing time, based on the last observed concentration for FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 72 h post-dose
Part 1: Clearance of FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 72 h post-dose
Part 1: AUC% extrapolated for FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 72 h post-dose
Part 2: Maximum plasma concentration of FDL169 (and metabolites) following multiple oral doses of FDL169 | Multiple points from pre-dose to 48 h post last dose
Part 2: Time to maximum plasma concentration of FDL169 (and metabolites) following multiple oral doses of FDL169 | Multiple points from pre-dose to 48 h post last dose
Part 2: Individual estimate of the terminal elimination rate constant of FDL169 (and metabolites) following multiple oral doses of FDL169 | Multiple points from pre-dose to 48 h post last dose
Part 2: Terminal half-life of FDL169 (and metabolites) following multiple oral doses of FDL169 | Multiple points from pre-dose to 48 h post last dose
Part 2: AUC from the time of dosing to the time of the last observed concentration for FDL169 (and metabolites) following multiple oral doses FDL169 | Multiple points from pre-dose to 48 h post last dose
Part 2: AUC extrapolated to infinity from dosing time, based on the last observed concentration for FDL169 (and metabolites) following multiple oral doses of FDL169 | Multiple points from pre-dose to 48 h post last dose
Part 2: Clearance of FDL169 (and metabolites) following multiple oral doses of FDL169 | Multiple points from pre-dose to 48 h post last dose
Part 2: AUC% extrapolated for FDL169 (and metabolites) following multiple oral doses of FDL169 | Multiple points from pre-dose to 48 h post last dose
Part 3: Maximum plasma concentration of FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 48 h post-dose
Part 3: Time to maximum plasma concentration of FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 48 h post-dose
Part 3: Individual estimate of the terminal elimination rate constant of FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 48 h post-dose
Part 3: Terminal half-life of FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 48 h post-dose
Part 3: AUC from the time of dosing to the time of the last observed concentration for FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 48 h post-dose
Part 3: AUC extrapolated to infinity from dosing time, based on the last observed concentration for FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 48 h post-dose
Part 3: Clearance of FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 48 h post-dose
Part 3: AUC% extrapolated for FDL169 (and metabolites) following single oral dose of FDL169 | Multiple points from pre-dose to 48 h post-dose

SECONDARY OUTCOMES:
Number of subjects with clinically significant changes in systolic and diastolic blood pressure following single and multiple oral doses of FDL169 | Multiple points from screening to follow-up (7 days after last dose)
Number of subjects with clinically significant changes in heart rate following single and multiple oral doses of FDL169 | Multiple points from screening to follow-up (7 days after last dose)
Number of subjects with clinically significant changes in oral temperature following single and multiple oral doses of FDL169 | Multiple points from screening to follow-up (7 days after last dose)
Number of subjects with clinically significant changes in oxygen saturation following single and multiple oral doses of FDL169 | Multiple points from screening to follow-up (7 days after last dose)
Number of subjects with clinically significant 12-lead ECG abnormalities following single and multiple oral doses of FDL169 | Multiple points from screening to follow-up (7 days after last dose)
Number of subjects with abnormal laboratory values following single and multiple oral doses of FDL169 | Multiple points from screening to follow-up (7 days after last dose)
Number of subjects experiencing treatment-related adverse events following single and multiple oral doses of FDL169 | Multiple points from screening to follow-up (7 days after last dose)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Elborn, MD, Principal Investigator — Queen's University
Locations (1):
- Celerion, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided